CLINICAL TRIAL: NCT03770546
Title: Amnion-Based Injections in the Shoulder for Adhesive Capsulitis and Osteoarthritis
Brief Title: Amnion-Based Injections in the Shoulder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure of institution to reach agreement with company supplying injections
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eugene Willis Brabston, Associate Professor, Orthopaedic Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300002242
Record Dates: First submitted 2018-11-21; First posted 2018-12-10 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis of the Shoulder; Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Osteoarthritis - Amnion Injection (Experimental): BioDRestore Elemental Tissue Matrix is a morselized, flowable tissue allograft derived from human amniotic tissues.
  Interventions: Biological: Amnion Injection
- Osteoarthritis - Betamethasone Injection (Active Comparator): Betamethasone Sodium Phosphate and Betamethasone Acetate injection (To clarify, this is one formulation/injected solution, not separate solutions/interventions)
  Interventions: Drug: Betamethasone injection
- Adhesive Capsulitis - Amnion Injection (Experimental): BioDRestore Elemental Tissue Matrix is a morselized, flowable tissue allograft derived from human amniotic tissues.
  Interventions: Biological: Amnion Injection
- Adhesive Capsulitis - Betamethasone Injection (Active Comparator): Betamethasone Sodium Phosphate and Betamethasone Acetate injection (To clarify, this is one formulation/injected solution, not separate solutions/interventions)
  Interventions: Drug: Betamethasone injection

INTERVENTIONS:
Biological: Amnion Injection — Per the manufacturer, this is considered an injection of tissue/organic matter.
  Arms: Adhesive Capsulitis - Amnion Injection; Osteoarthritis - Amnion Injection
Drug: Betamethasone injection — Routine steroid injection for these pathologies. Betamethasone Sodium Phosphate and Betamethasone Acetate injection.
  Arms: Adhesive Capsulitis - Betamethasone Injection; Osteoarthritis - Betamethasone Injection

SUMMARY:
Osteoarthritis (OA) of the shoulder is a common debilitating condition affecting up to 5% of the general population and as much as 32% of patients over 60 years of age. Clinically, OA is diagnosed by a combination of symptoms, such as slow onset of progressively worsening shoulder pain and stiffness over months to years (often with a history of minor trauma), and pain with activity. Physical exam may show tenderness and swelling, muscle atrophy, and decreased range of motion. Adhesive capsulitis (also called "Frozen Shoulder") is another common shoulder condition, affecting 2-5% of the general population. Frozen shoulder presents with a similar combination of symptoms, such as inability to sleep on the side of the affected shoulder, shoulder pain, and pain at extremes of active and passive range of motion.

Despite the ubiquitous nature of these conditions, various non-operative treatment modalities have been employed in their managements without a clearly superior alternative. The usual initial treatment strategy for both of these conditions is the same: a trial of conservative management. Conservative management includes physical therapy, supervised neglect, over-the-counter pain medications (including NSAIDs, like Advil), oral and intra-articular corticosteroid use (steroids), hydrodilatation (capsular distension to rupture), intra-articular hyaluronic acid injections. Despite several years of employing different modes of treatment, there is no evidence that places one treatment modality over the others, and patients will often need surgery.

Amniotic fluid's apparent ability to improve blood flow, re-organize collagen, and protect cartilage makes it theoretically ideal for disorders like osteoarthritis and frozen shoulder. In recent studies, it has shown efficacy in promoting ligament healing in the knee and promoting tendon and degenerative joint pain reduction and functional improvement. It has been useful as a material for cartilage repair when used as a scaffold. Intra-articular amnion membrane injection may have favorable outcomes in patients with osteoarthritis of the shoulder or frozen shoulder. To test this hypothesis, intra-articular amnion will be injected into the shoulders of 20 patients with moderate to severe osteoarthritis and 20 patients with frozen shoulder. The hypothesis is that improvement in short-term outcomes (pain, function, and range of motion) will be identified following amnion injection in these patients. The goal of this study is to lead to larger randomized controlled trials evaluating amnion against current forms of treatment for osteoarthritis.

DETAILED DESCRIPTION:
Amnion injections are commonly performed by community orthopaedic surgeons for many conditions, including osteoarthritis, rotator cuff tears, tendinitis, and others. Human placental tissue has been reported to contain biochemical and immunologic properties that play key roles in regulation of the inflammation-healing cycle. Amnion-chorion membrane has been shown to contain high concentrations of collagens, transforming growth factor beta suppressors, and inhibitors of matrix metalloproteinases that provide strong scaffolding, suppress scar formation, and regulate tissue remodeling, respectively. The amnion injection is a morselized, flowable tissue allograft derived from human amniotic tissues. The amniotic tissue comes from placenta, donated by pre-screened healthy women undergoing scheduled C-sections. It is processed into a form that can be injected.

Similarly, in a recent study injection of micronized dehydrated human amnion-chorion membrane slowed the development of cartilaginous lesions and led to a decreased number of erosions in a rat model of osteoarthritis. There is also an emerging body of literature investigating its use in osteoarthritis of the knee, with promising early results. In one study human amniotic suspension allograft was injected into patients with symptomatic knee osteoarthritis. No significant reactions were noted and the feasibility of injection for treatment of the osteoarthritis in the knee was demonstrated. Another study found that human amniotic fluid had a positive effect on tibia fracture healing through a rat model. In an osteoarthritis model, injection demonstrated attenuation of cartilage destruction and significant increases in cartilage thickness and volume. Finally, patients with plantar fasciitis noted significant improvement in symptoms, and American Orthopaedic Foot and Ankle Society Hindfoot scores (pain, function, alignment) compared to controls. These studies suggest the safety and efficacy of amnion-based injections in treating specific orthopaedic pathologies.

Osteoarthritis and adhesive capsulitis are two common pathologies of the shoulder. There is a variety of options for conservative management including physical therapy, pain medications, and injections, but no evidence that places one modality over another. The purpose of this study is the evaluate the effectiveness of amniotic fluid injection in treating these pathologies. In this study intra-articular amnion will be injected into the shoulders of patients with moderate to severe osteoarthritis and patients with frozen shoulder and assessing pain, function and range of motion over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Clinical diagnosis of adhesive capsulitis, clinically in the frozen phase at the time of enrollment OR Clinical diagnosis of osteoarthritis of the shoulder.
* Symptoms for 2-6 months
* Failure of conservative management.
* > 25% reduction in active range of motion in >= 2/3 planes of motion in the affected shoulder.
* No alternative medical explanation for symptoms

Exclusion Criteria:

* Alternative explanation for symptoms including neurological disorders, or like conditions
* Pregnancy or desire to become pregnant
* Discretion of the enrolling clinician

Exclusion in Amnion Injection Group:

• Intra-articular steroid injection within 6 months of enrollment or surgical intervention in the within 12 months of enrollment in affected shoulder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 0-12 months after injection
  Measured via goniometer
Strength | 0-12 months after injection
  Measured via dynamometer

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index for shoulder pain and function | 0-12 months after injection
  Patient reported outcome measure of shoulder pain and function. Score is between 0% and 100%. There are 5 questions in on the pain scale and 8 questions on the disability scale, each rated from 0-10. Pain score is the sum of the ratings of the 5 question out of 50 converted to a percentage (0-100%). Disability score is the sum of the ratings of the 8 questions out of 80 converted to a percentage (0-100%). The overall score is a sum of the ratings for all 13 questions out of 130 converted to a percentage (0-100%). A higher score indicates worse outcomes.
Short-Form Health Survey 36 for physical health, mental health, pain and limitation of activities | 0-12 months after injection
  Patient reported outcome measure of physical health, mental health, pain and limitation of activities. There is a physical health score and mental health score, each a number from 0-100. A higher score indicates better health.
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form of shoulder function | 0-12 months after injection
  Patient reported outcome measure assessing shoulder function with a score between 0 and 100. A higher score represents better shoulder function.
Simple Shoulder Test of shoulder function | 0-12 months after injection
  Patient reported outcome measure of shoulder function. It is a set of 12 yes/no questions. The score is calculated as the number of "yes" response out of 12 converted to a percentage (0-100%). A higher score represents better shoulder function.
Disabilities of the Arm, Shoulder, and Hand Questionnaire of arm, shoulder, and hand function | 0-12 months after injection
  Patient reported outcome measure assessing arm, shoulder, and hand function. This is a score ranging from 0-100 with a higher score indicating worse function of the upper extremities.
Visual Analog Scale for Pain | 0-12 months after injection
  Patient reported outcome measure assessing pain with a scale from 0-100, a higher score indicating greater pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bal A, Eksioglu E, Gulec B, Aydog E, Gurcay E, Cakci A. Effectiveness of corticosteroid injection in adhesive capsulitis. Clin Rehabil. 2008 Jun;22(6):503-12. doi: 10.1177/0269215508086179. PMID 18511530
- [Background] Carette S, Moffet H, Tardif J, Bessette L, Morin F, Fremont P, Bykerk V, Thorne C, Bell M, Bensen W, Blanchette C. Intraarticular corticosteroids, supervised physiotherapy, or a combination of the two in the treatment of adhesive capsulitis of the shoulder: a placebo-controlled trial. Arthritis Rheum. 2003 Mar;48(3):829-38. doi: 10.1002/art.10954. PMID 12632439
- [Background] Lorbach O, Anagnostakos K, Scherf C, Seil R, Kohn D, Pape D. Nonoperative management of adhesive capsulitis of the shoulder: oral cortisone application versus intra-articular cortisone injections. J Shoulder Elbow Surg. 2010 Mar;19(2):172-9. doi: 10.1016/j.jse.2009.06.013. Epub 2009 Oct 1. PMID 19800262
- [Background] Willett NJ, Thote T, Lin AS, Moran S, Raji Y, Sridaran S, Stevens HY, Guldberg RE. Intra-articular injection of micronized dehydrated human amnion/chorion membrane attenuates osteoarthritis development. Arthritis Res Ther. 2014 Feb 6;16(1):R47. doi: 10.1186/ar4476. PMID 24499554
- [Background] Vines JB, Aliprantis AO, Gomoll AH, Farr J. Cryopreserved Amniotic Suspension for the Treatment of Knee Osteoarthritis. J Knee Surg. 2016 Aug;29(6):443-50. doi: 10.1055/s-0035-1569481. Epub 2015 Dec 18. PMID 26683979
- [Background] Kerimoglu S, Livaoglu M, Sonmez B, Yulug E, Aynaci O, Topbas M, Yarar S. Effects of human amniotic fluid on fracture healing in rat tibia. J Surg Res. 2009 Apr;152(2):281-7. doi: 10.1016/j.jss.2008.02.028. Epub 2008 Mar 18. PMID 18499130
- [Background] Raines AL, Shih MS, Chua L, Su CW, Tseng SC, O'Connell J. Efficacy of Particulate Amniotic Membrane and Umbilical Cord Tissues in Attenuating Cartilage Destruction in an Osteoarthritis Model. Tissue Eng Part A. 2017 Jan;23(1-2):12-19. doi: 10.1089/ten.TEA.2016.0088. Epub 2016 Nov 18. PMID 27707109
- [Background] Zelen CM, Poka A, Andrews J. Prospective, randomized, blinded, comparative study of injectable micronized dehydrated amniotic/chorionic membrane allograft for plantar fasciitis--a feasibility study. Foot Ankle Int. 2013 Oct;34(10):1332-9. doi: 10.1177/1071100713502179. Epub 2013 Aug 14. PMID 23945520